CLINICAL TRIAL: NCT06900114
Title: Disease Burden Transition of Mucormycosis in Hematologic Malignancies Population Across Covid 19 Era: a Single-center Comparative Analysis From China
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2024056
Record Dates: First submitted 2024-11-29; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-11

CONDITIONS: Mucormycosis; Hematologic Malignancies; COVID-19
Keywords: Mucormycosis; Hematologic Malignancies; COVID-19; China
MeSH Terms: conditions — Mucormycosis; Hematologic Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Covid 19 group: Divide the patients into pre-covid 19 group(2015.01-2019.12) and covid 19 group(2020.1-2023.12) according to the time period.
- Covid 19 group: Divide the patients into pre-covid 19 group(2015.01-2019.12) and covid 19 group(2020.1-2023.12) according to the time period.

SUMMARY:
The project intends to carry out a retrospective study on the epidemiology, predisposing factors, clinical manifestations, diagnosis, treatment, prognosis and economic burden of mucormycosis in a Chinese single-center allogeneic hematopoietic stem cell transplantation population. The project was conducted at the Blood Diseases Hospital, Chinese Academy of Medical Sciences, which has rich experience in hematopoietic stem cell transplantation and has completed more than 3,000 cases of various types of HSCT, 400 allogeneic hematopoietic stem cell transplants per year, and routine bronchoscopy and application of guideline-recommended regimens for the treatment of mucormycosis. This study will objectively reflect the current management status of allogeneic hematopoietic stem cell transplantation combined with mucormycosis in Chinese transplant centers. Through systematic analysis of the changes in the management of mucormycosis in Chinese patients undergoing hematopoietic stem cell transplantation, to gain perspective into the impact of Covid19, diagnostic techniques, and new drugs on the incidence, diagnosis and treatment of mucormycosis . This will has a profound impact on optimizing the management strategies of mucormycosis in patients undergoing hematopoietic stem cell transplantation in the future.

DETAILED DESCRIPTION:
Divide the patients into pre-covid 19 group(2015.01-2019.12) and covid 19 group(2020.1-2023.12) according to the time period.

Objectives:

1.Conduct a comparative analysis in 2015-2020 stage (Pre-Covid Era) and 2020-2024 stage (Covid Era). To summarize and compare the characteristics of Mucormycosis in Chinese hematologic malignancies population from the aspects of incidence, mucorus species, types of mucormycosis, diagnostic techniques, treatment methods (surgical +drugs), pharmaceutical economics and prognosis between two stages. Objectively reflect the current management status of Mucormycosis in this population.

2 Analyze the possible causes of the epidemiology changing of mucormycosis: COVID19 influence, the advancement of diagnostic technology(NGS, respiratory endoscope intervention technique etc.) and other factors.

3 Impact of treatment progress on disease prognosis and burden: the status of surgery changes; To investigate the efficacy, safety and therapeutic status of posaconazole and other antifungal drugs in the treatment of Mucormycosis, and analyze the impact of the new antifungal drugs on the prognosis.

Data collection:

According to the information provided in the medical records and test results, enter the relevant data: including baseline characteristics, complications, clinical manifestations, laboratory tests, bronchoscopy results, imaging findings, fungal prophylaxis medication, therapeutic medication, surgical conditions and prognosis.

Results:

1. Incidence difference of invasive mucormycosis between two stages;
2. Risk factors difference of invasive mucormycosis between two stages;
3. Difference of Clinical types, imaging features and bronchoscopic features of invasive mucormycosis in hematologic malignancies between two stages;.
4. Changing of etiology and histopathological results of invasive mucormycosis in hematologic malignancies between two stages;.
5. History of antifungal drug exposure in hematologic malignancies patients with invasive mucormycosis;
6. Treatment regimen and course changing of invasive mucormycosis
7. Prognosis of invasive mucormycosis in hematologic malignancies patients;
8. Economic burden transition of invasive mucormycosis in hematologic malignancies patients including average length of hospital stay, cost of antifungal therapy etc.
9. Incidence and characteristics of invasive pulmonary mucormycosis in allogeneic hematopoietic stem cell transplantation patients during two stages.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematologic diseases who undergoes hematopoietic stem cell transplantation in the center from January 2015 to December 2023.
2. Age≥18 years old.
3. Patients who were diagnosed with mucormycosis(proven or probable) in accordance with the 2008 EORTC/MSG criteria and Revised EORTC/MSGERC 2020 Criteria.[8][9].
4. The patients themselves or their authorized clients agree to participate in the clinical study and sign the informed consent.

Exclusion Criteria:

1. Patients with fungal infections other than mucormycosis were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with mucormycosis(proven or probable) in accordance with the 2008 EORTC/MSG criteria and Revised EORTC/MSGERC 2020 Criteria.
  Mucormycosis is a rare opportunistic fungal infection typically characterized by rapid progression, the main susceptible population is patients with diabetes and severe underlying diseases of immunocompromised patients with poor glycemic control (e.g., hematologic malignancies, hematopoietic stem cell transplantation, solid organ transplantation, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To summarize and compare the characteristics of Mucormycosis in Chinese hematologic malignancies population | 2 YEARS
  Conduct a comparative analysis in 2015-2020 stage (Pre-Covid Era) and 2020-2024 stage (Covid Era). To summarize and compare the characteristics of Mucormycosis in Chinese hematologic malignancies population from the aspects of incidence, mucorus species, types of mucormycosis, diagnostic techniques, treatment methods (surgical +drugs), pharmaceutical economics and prognosis between two stages. Objectively reflect the current management status of Mucormycosis in this population.

SECONDARY OUTCOMES:
Analyze the possible causes of the epidemiology changing of mucormycosis: COVID19 influence, the advancement of diagnostic technology(NGS, respiratory endoscope intervention technique etc.) and other factors. | 2 YEARS
  Analyze the possible causes of the epidemiology changing of mucormycosis: COVID19 influence, the advancement of diagnostic technology(NGS, respiratory endoscope intervention technique etc.) and other factors.
Impact of treatment progress on disease prognosis and burden: the status of surgery changes | 2 YEARS
  Impact of treatment progress on disease prognosis and burden: the status of surgery changes; To investigate the efficacy, safety and therapeutic status of posaconazole and other antifungal drugs in the treatment of Mucormycosis, and analyze the impact of the new antifungal drugs on the prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China